CLINICAL TRIAL: NCT00861731
Title: The Metabolic and Anti-Inflammatory Effects of Combined Ezetimibe and Simvastin Therapy, as Compared to Simvastatin Alone, in Patients With Chronic Proteinuric Nephropathy
Brief Title: Ezetimibe/Simvastatin Combination in Proteinuric Nephropathy
Acronym: VICTORY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliero Universitaria di Sassari (Other)
Responsible Party: Andrea Ercole Satta, Istituto di Patologia Speciale Medica e Metodologia Clinica - AOU di Sassari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOUSS-Nefologia-001
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Hypercholesterolemia; Chronic Nephropathy
Keywords: chronic renal failure; proteinuria; apolipoprotein; c reactive protein
MeSH Terms: conditions — Hypercholesterolemia; Kidney Failure, Chronic; Proteinuria | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): hypolipidemic treatment
  Interventions: Drug: simvastatin
- 2 (Sham Comparator): hypolipidemic treatment
  Interventions: Drug: EZE/simvastatin
- 3 (Sham Comparator): hypolipidemic treatment
  Interventions: Drug: EZE/simvastatin

INTERVENTIONS:
Drug: simvastatin — simvasatin therapy alone at the dose of 40 mg/day
  Arms: 1
Drug: EZE/simvastatin — EZE/simvastatin combined therapy at the dose of 10/20 mg/day
  Arms: 2
Drug: EZE/simvastatin — EZE/simvastatin combined therapy at the dose of 10/40 mg/day
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether, in patients with chronic proteinuric nephropathy and dyslipidemia, ezetimibe-simvastatin combined therapy is more effective than statin alone to achieve the optimum lipid control, and if this translates to an improvement of the markers of vascular damage. Thirty hypertensive patients in stable therapy with RAS inhibitors, with low-density lipoprotein (LDL) cholesterol superior to 100 mg/ml, are treated with three different hypolipidemic regimens: Simvastatin alone (40 mg/day) or ezetimibe/simvastatin combined therapy (10/20 or 10/40 mg/day).

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) have an increased incidence of cardiovascular morbidity and mortality. Presence of hypertension, lipid abnormalities and inflammation each contribute to increased cardiovascular risk. Therefore blood pressure control slows the progression of CKD towards End Stage Renal Failure (ESRF) improving clinical outcome.

Instead the contribution of lipid abnormalities is still not completely understood, mainly because dyslipidemia interferes with a number of non-traditional cardiovascular risk factors, particularly the activated acute-phase response.

In proteinuric patients, dyslipidemia has a highly atherogenic profile, with increased total and low-density lipoprotein (LDL) cholesterol, triglyceride, and lipoprotein(a) serum levels, as well as decreased HDL cholesterol. Numerous studies have indicated that treatment of dyslipidemia with a statin decreases cardiovascular morbidity and mortality. Experimental and clinical evidences show that statin, in addition to ameliorate lipid profile, may have specific renoprotective properties and, combined to Renin-Angiotensin System (RAS) inhibitor therapy, may synergize their antiproteinuric effects.

Preliminary data are also available data that the combination of statin to ezetimibe (EZE), a cholesterol absorption inhibitor, produces an additional decrease in LDL cholesterol and C-reactive protein levels, over that achieved with statin monotherapy.

Thus, adding the potential antinflammatory effect to hypolipidemic efficacy, combined therapy may expand the renal and cardioprotective potentiality. It may also permit a reduction of statin therapeutic dose improving safety profile. Therefore EZE-statin combination therapy may be an effective therapeutic option to statin alone in patients with high cardiovascular risk, such as chronic proteinuric patients.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* LDL-cholesterol > 100 mg/dl (without concomitant hypolipidemic drugs) in patients whit high cardiovarscular risk for the concomitant presence of:
* proteinuric chronic nephropathy defined as creatinine clearance > 20 ml/min/1,73 m2 combined to a urinary protein excretion rate > 0,3 g/24h, without evidence of urinary tract infection or overt heart failure (New York Heart Association class III or more)
* hypertension defined as a systolic or diastolic blood pressure > 140 or 90 mmHg respectively (or less in patients with concomitant antihypertensive therapy)

Exclusion Criteria:

* previous or concomitant treatment with steroids, anti-inflammatory and immunosuppressive agents
* evidence or suspicion of renovascular disease, obstructive uropathy, type I diabetes mellitus, vasculitides, history of poor tolerance or allergy to ACEi and ATA, statin or EZE, drug abuse or pregnancy
* inability to fully understand the purposes/risks of the study and to provide a written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
To assess whether EZE-statin combined therapy is more effective than statin alone to achieve the optimum lipid control (LDL-cholesterol < 70 mg/dl) in chronic proteinuric nephropathy. | at baseline and every 4 months after therapy start

SECONDARY OUTCOMES:
To assess the effect of EZE-statin combined therapy vs statin monotherapy on other outcome variables including: - renal parameters - inflammatory status - markers of endothelial dysfunction | after one year observational period

CONTACTS AND LOCATIONS:
Overall Officials: Andrea E Satta, MD, Principal Investigator — Istituto di Patologia Medica -Azienda Ospedaliero Universitaria di Sassari
Locations (1):
- Istituto di Patologia Medica - Azienda Ospedaliero Universitaria, Sassari, Italy

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Zinellu A, Sotgia S, Sotgiu E, Assaretti S, Baralla A, Mangoni AA, Satta AE, Carru C. Cholesterol lowering treatment restores blood global DNA methylation in chronic kidney disease (CKD) patients. Nutr Metab Cardiovasc Dis. 2017 Sep;27(9):822-829. doi: 10.1016/j.numecd.2017.06.011. Epub 2017 Jun 28. PMID 28755807